CLINICAL TRIAL: NCT03928314
Title: An Open-label Phase 1b Study of ORIC-101 in Combination With Anticancer Therapy in Patients With Advanced or Metastatic Solid Tumors
Brief Title: Study of ORIC-101 in Combination With Anticancer Therapy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: IND Withdrawn
Sponsor: ORIC Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 101-18101
Record Dates: First submitted 2019-04-19; First posted 2019-04-26 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Solid Tumor
Keywords: GR antagonist; Glucocorticoid receptor antagonist
MeSH Terms: interventions — 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Intervention Model Description: Standard 3+3 dose escalation design, followed by dose expansion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (Part I) (Experimental): ORIC-101 dosed orally, once per day, for 5 or 7 days/week in combination with nab-paclitaxel (75 or 100 mg/m2 on Days 1, 8, and 15) of each 28-day cycle.
  Interventions: Drug: ORIC-101; Drug: Nab-paclitaxel
- Dose Expansion (Part II) (Experimental): RP2D dose
  Interventions: Drug: ORIC-101; Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: ORIC-101 — ORIC-101 once daily, 5 or 7 days/week, for 21 days of each 28-day cycle
Drug: Nab-paclitaxel — 75 or 100 mg/m2 Days 1, 8, and 15 of each 28-day cycle

SUMMARY:
The purpose of this study is to establish the recommended Phase 2 dose (RP2D), safety, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary antitumor activity of ORIC-101 in combination with nab-paclitaxel or other anticancer therapies when administered to patients with advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
ORIC-101 is a small molecule GR antagonist being developed for the treatment of patients with solid tumor malignancies. Mechanistically, ORIC-101 inhibits GR transcriptional activity and blocks the pro-survival signals mediated by the activated nuclear receptor.

This is an open-label, uncontrolled, multicenter, dose-finding study to assess the safety and preliminary antitumor activity of ORIC-101 in combination with nab-paclitaxel or other anticancer therapy in patients with advanced or metastatic solid tumors. The study will begin with dose finding in combination initially with nab-paclitaxel in patients with various solid tumors (Part I); additional dose expansion cohorts in specific tumor types with nab-paclitaxel (Part II) or with other anticancer therapies may be evaluated through protocol amendment(s).

The study will first evaluate intermittent administration (5 days on, 2 days off for 21 days) of ORIC-101 followed by continuous administration (daily for 21 days) in combination with nab-paclitaxel using a standard 3+3 dose escalation design.

In Part II, patients will be enrolled across four cohorts of advanced or metastatic disease:

* pancreatic ductal adenocarcinoma (PDAC)
* ovarian cancer
* triple negative breast cancer (TNBC)
* other solid tumors

ELIGIBILITY:
Inclusion Criteria (Part I):

* Advanced or metastatic solid tumor, with the exception of neuroendocrine tumors that secrete adrenocorticotropic hormone (ACTH) or corticotropin-releasing hormone (CRH), for which no alternative effective standard therapy is available or for which standard therapy is considered unsuitable or intolerable
* Measurable disease (ie, presenting with at least one measurable lesion per RECIST 1.1)
* Radiographic evidence of a lesion that may be safely biopsied by core needle biopsy
* For patients with treated, stable CNS metastases that are asymptomatic: no evidence of progression for at least 4 weeks after CNS-directed treatment as determined by clinical examination and brain imaging. Patients must not require steroids
* ECOG performance status 0 or 1
* Life expectancy of at least 3 months
* Available archival FFPE tissue for submission to central laboratory
* Male: must agree to birth control requirements and Female: not pregnant, breastfeeding, and meets requirements regarding women of child-bearing potential
* Capable of giving signed informed consent
* Agreement and ability to undergo two on-study biopsies, as follows, through a procedure that is deemed to be clinically feasible and not carry significant risk:

  * one pre-treatment tumor biopsy obtained prior to dosing; and
  * one post-treatment tumor biopsy during Cycle 2

Exclusion Criteria (Part I):

* Any other current or active malignancy
* Grade 2 or higher peripheral neuropathy
* Known human immunodeficiency virus (HIV) infection
* Major surgery within 21 days prior to Cycle 1 Day 1 or incomplete recovery from adverse effects resulting from such procedure
* Females: history of unexplained vaginal bleeding in the 8 weeks prior to planned study treatment
* History of Cushing's syndrome or adrenal insufficiency
* Other concurrent serious uncontrolled medical, psychological, or addictive conditions that may interfere with planned study treatment or adherence to protocol
* Prior or current treatment with ORIC-101 or any other GR antagonist (eg, mifepristone, relacorilant)
* Current or requirement for chronic use of systemic corticosteroids with the exception of inhaled, topical, intraocular, intranasal, or intraarticular corticosteroids.
* Current or expected on-study treatment with specified strong CYP3A4 inhibitors or inducers
* Treatment with another investigational medicinal product (within 3 weeks prior to starting study treatment)
* Receiving any other anticancer therapy, radiotherapy, or herbal (alternative) medicines within 7 days prior to starting study treatment
* Use of hormone replacement therapy by females
* Current enrollment in any other therapeutic clinical study involving an investigational study treatment
* Presence of Hepatitis B surface antigen at screening
* Positive Hepatitis C antibody test result at screening or within 3 months prior to starting study treatment
* Positive Hepatitis C RNA test result at screening or within 3 months prior to first dose of study treatment
* Unacceptable laboratory criteria:

  * ANC <1500 cells/mm3 (1.5 × 103 cells/mm3)
  * Platelets <100,000 /µL (100 × 109 /L)
  * Hemoglobin <9.0 g/dL (90 g/L)
  * Albumin <3.0 g/dL (30 g/L)
  * AST (SGOT) or ALT(SGPT) >2.5 × ULN
  * AST (SGOT) or ALT (SGPT) >2.5 and ≤5.0 × ULN is acceptable for patients with liver metastases
* Bilirubin >1.5 × ULN:

  * Isolated bilirubin >1.5 × ULN is acceptable if bilirubin is fractionated and direct bilirubin <35% of total bilirubin
  * Bilirubin >1.5 and ≤3.0 × ULN is acceptable for patients with known Gilbert's disease
* QTcF >450 msec for males; QTcF >470 msec for females; or QTcF >480 msec for those with bundle branch block (BBB)
* Consumption of Seville oranges, grapefruit or grapefruit juice, pomelos, exotic citrus fruits, grapefruit hybrids, or fruit juices containing these fruits from 10 days before the start of study treatment
* Sensitivity to any of the study treatments, or components thereof, or drug or other allergy that, in the opinion of the investigator, contraindicates participation in the study.
* Any other condition or circumstance (eg, familial, sociological, inability to swallow oral study drug) that, in the opinion of the investigator, may interfere with protocol compliance or contraindicates participation in the study.

Expansion Cohorts Part II Inclusion Criteria:

* PDAC: Advanced or metastatic PDAC previously treated with and progressed on a fluoropyrimidine-based regimen and a taxane-containing chemotherapy regimen (eg, gemcitabine + nab-paclitaxel). Pancreatic neuroendocrine tumors, lymphoma of the pancreas, acinar pancreatic cancer, or ampullary cancer are not eligible.
* Ovarian Cancer: Advanced or metastatic high grade serous or endometrioid epithelial ovarian, primary peritoneal, fallopian tube cancer or ovarian carcinosarcoma, previously treated with and progressed on a taxane-containing chemotherapy regimen; clear cell, mucinous and borderline histologic subtypes are not eligible; must have received at least one line of therapy with evidence of cancer progression within 6 months after the last dose of platinum-based therapy (ie, having a platinum-free interval of <6 months [platinum resistant]), or progressive disease during or immediately after primary platinum-therapy, (ie, platinum refractory).
* TNBC: Advanced or metastatic ER-negative, PR-negative, HER2-negative primary breast cancer previously treated and progressed on a taxane-based chemotherapy regimen; no previous or synchronous second breast cancer, unless also confirmed ER-, PR- and HER2-negative; must have received at least one line of therapy in the metastatic setting.
* Other Solid Tumor: Other advanced or metastatic solid tumor previously treated with and progressed on a taxane-based chemotherapy regimen, with the exception of metastatic colorectal cancer, primary brain tumors, and neuroendocrine tumors that secrete ACTH or CRH; must have received no more than 4 prior lines of cytotoxic or myelosuppressive therapy

Other Key Inclusion Criteria:

* At least 18 years of age
* ECOG performance status 0 or 1
* Measurable disease as assessed centrally using RECIST 1.1
* Treated, stable CNS metastases must be asymptomatic and must not require steroids
* Agreement and ability to undergo two on-study biopsies, one pre-treatment obtained prior to dosing and during Cycle 2
* Adequate organ function as defined by the following criteria:

  * ANC ≥1500 cells/mm3 (1.5 × 103 cells/mm3)
  * Platelets ≥100,000 /µL (100 × 109 /L)
  * Hemoglobin ≥9.0 g/dL (90 g/L)
  * Albumin ≥3.0 g/dL
  * AST (SGOT) or ALT (SGPT) ≤2.5 × ULN, ≤5.0 × ULN for patients with liver metastases
  * Bilirubin ≤1.5 × ULN; patients with a known history of Gilbert's syndrome and/or isolated elevations of indirect bilirubin are eligible
  * QTcF ≤480 msec
* Ability to swallow ORIC-101 intact without chewing or crushing the capsules or tablets
* Adequate gastrointestinal absorption. If the patient has undergone gastric bypass surgery and/or surgery of gastrointestinal or hepatobiliary tract, the patient must demonstrate adequate absorption as evidenced by albumin ≥3.0 g/dL, controlled pancreatic insufficiency (if present), and lack of evidence of malabsorption

Expansion Cohorts Part II Exclusion Criteria:

* Any other current or active malignancy
* Prior or current treatment with ORIC-101 or any other GR antagonist (eg, mifepristone, relacorilant)
* Concurrent treatment with any other anticancer therapy including chemotherapy, hormonal therapy, immunotherapy, radiotherapy, chemoembolization, targeted therapy, or an investigational agent within 28 days prior to Cycle 1 Day 1
* Major surgery or radiotherapy within 21 days prior to Cycle 1 Day 1 or incomplete recovery from adverse effects resulting from such procedures; palliative radiotherapy within 1 week of Cycle 1 Day 1
* Systemic, inhaled, or prescription strength topical corticosteroids within 21 days prior to Cycle 1 Day 1; short courses (≤5 days) for non-cancer-related reasons are allowed if clinically required
* Grade 2 (moderate) or higher peripheral neuropathy per CTCAE v5.0; patients with mild peripheral neuropathy may be eligible at the discretion of the investigator in consultation with ORIC
* All other toxicities from prior therapy (except alopecia) that have not resolved to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0 ≤ Grade 1
* Females: history of unexplained vaginal bleeding in the 8 weeks prior to Cycle 1 Day 1 (given potential for ORIC-101 to exacerbate such bleeding)
* Females: use of hormone replacement therapy; hormone replacement therapy must be discontinued to allow for confirmation of postmenopausal status
* History of Cushing's syndrome or adrenal insufficiency
* Current (within 10 days prior to Cycle 1 Day 1) or expected on-study treatment with specified strong CYP3A4 inhibitors or inducers
* Known human immunodeficiency virus (HIV) infection, unless patient is healthy and has a low risk of AIDS-related outcomes
* Presence of Hepatitis B surface antigen (HBsAg) at screening
* Positive Hepatitis C (HCVAb) antibody test result at screening or within 3 months prior to Cycle 1 Day 1. NOTE: Patients with positive HCVAb due to prior resolved disease can be enrolled if a confirmatory negative Hepatitis C RNA test is obtained
* Positive Hepatitis C RNA test result at screening or within 3 months prior to Cycle 1 Day 1. NOTE: Test is optional and patients with negative HCVAb test are not required to also undergo Hepatitis C RNA testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2022-09-22 (Actual); Study Completion 2023-12-04 (Actual)

PRIMARY OUTCOMES:
Part I: Recommended Phase 2 Dose (RP2D) | 12 months
  RP2D as determined by 3+3 dose escalation design
Part II: Objective Response Rate (ORR) | 18 months
  Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and assessed by Blinded Independent Central Review (BICR)

SECONDARY OUTCOMES:
Part I: Maximum plasma concentration (Cmax) | 28 Days
  PK of ORIC-101 in combination with nab-paclitaxel
Part I: Time of maximum observed concentration (Tmax) | 28 Days
  PK of ORIC-101 in combination with nab-paclitaxel
Part I: Area under the curve (AUC(0-t)) | 28 Days
  PK of ORIC-101 in combination with nab-paclitaxel
Parts I and II: Number of Participants with Adverse Events | 36 months
  Safety and tolerability of ORIC-101 in combination with nab-paclitaxel
Parts I and II: Number of Participants with Abnormal Laboratory Values | 36 months
  Safety and tolerability of ORIC-101 in combination with nab-paclitaxel
Parts I and II: Number of Participants with Abnormal 12-lead ECG | 36 months
  Safety and tolerability of ORIC-101 in combination with nab-paclitaxel
Parts I and II: Number of Participants with Abnormal Vital Signs | 36 months
  Safety and tolerability of ORIC-101 in combination with nab-paclitaxel
Part I: Number of Participants with Antitumor Activity | 36 months
  Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria
Part II: Duration of Response (DOR) | 36 months
  Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and assessed by Blinded Independent Central Review (BICR)
Part II: Progression-Free Survival (PFS) | 36 months
  Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and assessed by Blinded Independent Central Review (BICR)
Part II: Overall Survival (OS) | 36 months
  Time from first dose of ORIC-101 in combination with nab-paclitaxel to death
Part II: Investigator-assessed ORR | 36 months
  Response Evaluation Criteria in Solid Tumors (RECIST) 1.1

OTHER OUTCOMES:
Parts I and II: Number of Participants with GR Expression by IHC | 36 months
  Level of GR expression by IHC in tumor tissue samples

CONTACTS AND LOCATIONS:
Overall Officials: Pratik S. Multani, MD, Study Director — ORIC Pharmaceuticals
Locations (12):
- United States (12):
  - Stanford Cancer Institute, Palo Alto, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - University of Colorado - PPDS, Aurora, Colorado
  - Florida Cancer Specialists & Research Institute, Lake Mary, Florida
  - Florida Cancer Specialists & Research Institute, Sarasota, Florida
  - Oregon Health & Science University, Portland, Oregon
  - Tennessee Oncology NASH - SCRI - PPDS, Nashville, Tennessee
  - Mary Crowley Cancer Research Centers - Medical City, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology, San Antonio, Texas
  - University of Utah - Huntsman Cancer Institute - PPDS, Salt Lake City, Utah
  - Virginia Cancer Specialists, PC, Fairfax, Virginia

REFERENCES:
- [Derived] Chen CT, Khanna V, Kummar S, Abdul-Karim RM, Sommerhalder D, Tolcher AW, Ueno NT, Davis SL, Orr DW, Hamilton E, Patel MR, Spira AI, Jauhari S, Florou V, Duff M, Xu R, Wang J, Barkund SR, Zhou H, Pankov A, Kong W, Jahchan NS, Jackson EL, Sun JD, Junttila MR, Multani PS, Daemen A, Chow Maneval E, Munster PN. ORIC-101, a Glucocorticoid Receptor Antagonist, in Combination with Nab-Paclitaxel in Patients with Advanced Solid Tumors. Cancer Res Commun. 2024 Sep 1;4(9):2415-2426. doi: 10.1158/2767-9764.CRC-24-0115. PMID 39177285